CLINICAL TRIAL: NCT06010537
Title: A Single-center, Randomized, Open-label, Single-dose Study of Polysaccharide Superparamagnetic Iron Oxide Injection in Healthy Subjects to Evaluate Magnetic Resonance Imaging in Multiple Dose Groups
Brief Title: Contrast-enhanced Magnetic Resonance Imaging With Polysaccharide Superparamagnetic Iron Oxide Nanoparticle
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: YHT-I-03
Record Dates: First submitted 2023-08-20; First posted 2023-08-24 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- polyglucose superparamagnetic iron oxide injection 2.5 mg/kg (Experimental): Intravenous injected polysaccharide superparamagnetic iron oxide injection at 2.5 mg/kg dose;
  Interventions: Drug: polysaccharide superparamagnetic iron oxide injection
- polyglucose superparamagnetic iron oxide injection 3.0 mg/kg (Experimental): Intravenous injected polysaccharide superparamagnetic iron oxide injection at 3.0 mg/kg dose;
  Interventions: Drug: polysaccharide superparamagnetic iron oxide injection

INTERVENTIONS:
Drug: polysaccharide superparamagnetic iron oxide injection — Polysaccharide superparamagnetic iron oxide injection is a magnetic resonance contrast agent.

SUMMARY:
This is a contrast-enhanced magnetic resonance imaging (MRI) study conducted on a single-administration of polyglucose superparamagnetic iron oxide injection. Two dose groups are set up in this study, 2.5 mg/kg and 3 mg/kg, and two subjects in each group received the test drug for safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Signing the informed consent form before the trial and fully understanding the content, process and possible adverse effects of the trial;
* Be able to complete the study according to the requirements of the trial protocol;
* Male subjects aged 18 to 40 years old (including the threshold);
* Subjects weighing no less than 50 kilograms. Body mass index (BMI) = weight (kg)/height2 (m2), BMI within the range of 19~26 (including the critical value);
* Health status: no mental abnormality, no history of cardiovascular system, nervous system, respiratory system, digestive system, urinary system, endocrine system and metabolic abnormalities;
* Vital signs, physical examination, laboratory tests, electrocardiogram and imaging tests are normal or abnormal without clinical significance;
* No pregnancy and voluntary use of effective contraception for at least 6 months from 2 weeks prior to dosing to the last use of the study drug.

Exclusion Criteria:

* Previously suffered from neuropsychiatric, respiratory, cardiovascular, gastrointestinal, hematologic-lymphatic, hepatic or renal insufficiency, endocrine, or musculoskeletal disorders, or other diseases, and in the judgment of the investigator, the previous medical history may have an impact on the magnetic resonance imaging procedure, the quality of the images, or the safety of the subject;
* Subjects with internal metal foreign bodies (dentures, contraceptive rings, metal implants, metal clips, etc.) and persons who are claustrophobic;
* Those who are allergic to the study drug, its metabolites or its excipients;
* Subjects who have smoked more than 5 cigarettes per day for 3 months prior to the trial;
* History of drug and/or alcohol abuse (14 units of alcohol per week: 1 unit = 360 ml of beer or 45 ml of spirits of 40% alcohol or 150 ml of wine);
* Blood donation or significant blood loss (> 450 ml) within 2 months prior to dosing;
* Use of any drug that alters liver enzyme activity (e.g., liver enzyme inhibitors chlorpromazine, cimetidine, ciprofloxacin, metronidazole, etc.; liver enzyme inducers barbiturates, carbamazepine, rifampicin, dexamethasone, etc.) in the 28 days prior to dosing;
* Use of any prescription medication, over-the-counter medication, any vitamin product or herbal remedy within 14 days prior to dosing;
* The need to use tobacco, alcohol and caffeinated beverages, or certain foods that may affect metabolism (e.g., grapefruit, grapefruit juice, etc.) during the trial period, or a significant change in dietary or exercise habits prior to the trial, or any other factor that affects the absorption, distribution, metabolism, or excretion of the drug;
* Use of an investigational drug or participation in a clinical trial of a drug within 2 months prior to dosing;
* Screening positive for hepatitis (including hepatitis B and C) and for AIDS and syphilis;
* Screening positive for drugs or a history of drug abuse within the past 5 years or drug use within the 3 months prior to the trial;
* Persons who have difficulty with MRI scanning or who cannot tolerate MRI scanning;
* Acute illness occurring during the pre-study screening phase or prior to study drug administration;
* Subjects who are unable or incapable of complying with ward regulations.
* The subject is unable to complete the trial for personal reasons.
* Other circumstances which, in the judgment of the investigator, make enrollment in the study unsuitable.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Adverse event rate | Baseline up to 144 hours
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).

SECONDARY OUTCOMES:
Contrast-enhanced magnetic resonance angiography (CE-MRA) | Before administration, 5 minutes, 12 hours, 24 hours, 36 hours, 48 hours after administration.
  CE-MRA of the whole heart and large arteries, coronary angiography and contrast-enhanced scan of the upper abdomen, the aorta and its main branches (left and right renal arteries, celiac trunk, superior mesenteric arteries, bilateral iliac arteries) as well as bilateral femoral arteries of the lower limbs will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Xinxiang Central Hospital, Xinxiang, Henan, China